CLINICAL TRIAL: NCT00951431
Title: Effect of Proton Pump Inhibitor on Gastric Emptying and Satiety Function in Patients With Functional Dyspepsia
Brief Title: Gastric Functions & Proton Pump Inhibitor( PPI) Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Justin Che-Yuen Wu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GFP
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Functional Dyspepsia
Keywords: Functional dyspepsia; PPI; postprandial fullness; delayed gastric emptying
MeSH Terms: conditions — Gastroparesis | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PPI (Experimental)
  Interventions: Drug: Esomeprazole
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esomeprazole — Esomeprazole 20mg daily for 8 weeks
  Other Names: Nexium
  Arms: PPI
Drug: Placebo — Placebo in the form of study drug
  Arms: Control

SUMMARY:
Functional dyspepsia is one of the most common digestive disorders. The pathophysiology of functional dyspepsia is uncertain. Proton pump inhibitor (PPI) has been recommended as the first line treatment for functional dyspepsia. However, the mechanism of symptom relief is unclear. Most of the previous studies were performed on healthy volunteers who received only a very short course of PPI. The correlation between symptom and gastric emptying is lacking in these studies.

Demographic data and anthropometric measurements will be obtained for baseline assessment. Patients are required to complete FGI Screening Questionnaire, Functional dyspepsia symptom questionnaire, gastroesophageal reflux disease (GERD) symptom questionnaire and irritable bowel syndrome (IBS) symptom questionnaire to have a thorough assessment of their GI symptoms. (1) Satiety test and ghrelin profile, and (2)gastric emptying test will be arranged as two individual visits.

After baseline investigations, patients will be randomly assigned to either Nexium 20 mg daily or identical looking placebo for 8 weeks. The patients will report their individual dyspeptic symptoms on weekly basis using a self-administered symptom questionnaire.

Satiety test and ghrelin profile, gastric emptying study will be repeated at the end of 8-week treatment.

Hypothesis: Long-term PPI relieves dyspeptic symptom through acceleration of gastric emptying rate.

DETAILED DESCRIPTION:
Background

Functional dyspepsia is one of the commonest digestive disorders. It is a functional gastrointestinal disorder which is characterized by chronic recurrent epigastric symptoms such as pain, burning and a variety of postprandial symptoms with absence of demonstrable organic pathology identified on investigations. It has been reported that functional dyspepsia affects 10-30% of adult population.

The pathophysiology of functional dyspepsia is uncertain. It is thought to be a heterogeneous disorder. Various factors have been implicated in the pathophysiology of functional dyspepsia. It has been reported that delayed gastric emptying, impaired proximal gastric accommodation, visceral hypersensitivity and Helicobacter pylori gastritis play a role in development of functional dyspepsia. However, the correlation between these physiological abnormalities and symptomatology of functional dyspepsia is poor. It is still controversial whether these pathophysiological factors are responsible for specific symptoms in functional dyspepsia.

While mechanism of functional dyspepsia is unclear, treatment has also been far from satisfactory. Proton pump inhibitor has been recommended as the first line treatment for functional dyspepsia and it has been shown that the use of PPI is associated with a 14% reduction in risk of persistent dyspepsia compared to placebo. However, the mechanism of symptom relief is unclear. While PPI exerts its effect primarily through suppression of acid-induced symptoms, recent studies have shown that PPI may affect gastric motility function such as gastric volume, gastric emptying and trigger of migratory motor complex. Most of these studies were performed on healthy volunteers who received only a very short course of PPI. The correlation between symptom and gastric emptying is lacking in these studies.

Aims

* To evaluate the effect of esomeprazole on gastric emptying
* To evaluate the relationship between dyspeptic symptom and gastric emptying

Hypothesis

Long-term PPI relieves dyspeptic symptom through acceleration of gastric emptying rate

Study design

Double-blind randomized placebo-controlled trial

Baseline assessment

* Demographic: age, gender
* Anthropometric measurements: body mass index, height, weight and waist circumference
* FGI Screening Questionnaire (v.2, 20090106) for screening of functional gastrointestinal disorder according to Rome III criteria.
* Functional dyspepsia symptom questionnaire (FDSQ) (20080416): an 8-item dyspeptic symptom score questionnaire: 4-point Likert scale for assessment of epigastric pain, epigastric burning, belching, bloating, postprandial fullness, early satiation, nausea and vomiting and a global dyspeptic symptom assessment.
* GERD Symptom questionnaire (GERDSQ) (20080416): GERD symptom score questionnaire.
* Irritable Bowel Syndrome Symptom questionnaire (IBSSQ) (20080428): IBS symptom score questionnaire.

Satiety test and ghrelin profile

After an overnight fast, the patients are instructed to ingest Ensure® (1.06 kcal/ml; 22% fat, 64% carbohydrate, and 14% protein) at constant rate of 30ml/min, and complete a Fullness Rating Scale (FRS) at 3-min intervals (ie. 0min, 3min, 6min…). The test will stop when a score of 4, which is equivalent to unbearable fullness, is reached in FRS. The volume (calorie) of Ensure that is ingested will be recorded and it serves as surrogate marker of satiety function. Serial blood sample (2ml each) will also be taken at 0, 30, 60, 90, 120min during test for assay of ghrelin and gastrin profile. If the test is stopped before 120 minutes, the remaining blood will still be taken according to schedule.

Gastric emptying test with FANci2

Measurement of gastric emptying rate of solid meal will be accomplished using 13C-octanoic acid breath test within 7 days after satiety test. After 12-hour fasting, the patient is required to ingest a pan-fried egg with 2 pieces of bread that contains 100 ul of 13C-octanoic acid dissolved in egg yolk. The exhaled gas will be collected at 15-minute intervals until 4 hours have passed. The 13CO2 content of the exhaled gas will be measured by a breath test device (FANci2, FAN GmbH.,Germany). 13CO2 is released after the 13C-octanoic acid enriched meal is emptied into the stomach and digested in duodenum.

Randomization of treatment

After baseline investigations, patients will be randomly assigned to either Esomeprazole 20 mg daily or identical looking placebo for 8 weeks. The random allocation sequence will be obtained from a computer-generated list of random numbers in blocks of 10. Concealed allocation is achieved by an independent staff who assigns treatments according to consecutive numbers in sealed envelopes. Study medications are dispensed as sealed packages in consecutive numbers. Medication adherence is measured by pill counts during interval visits.

Follow-up assessment

The patients will report their individual dyspeptic symptoms on weekly basis using a self-administered symptom questionnaire. At week 4 and week 8, they will need to give an additional rating on their overall symptom response using global symptom assessment. The patients are required to give a dichotomous response of either "yes" or "no" to the question stating "Do you have adequate relief of symptoms over the past 7 days?". Satiety test and blood sampling, gastric emptying study will be repeated at the end of 8-week treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with functional dyspepsia that fulfill Rome III criteria attending GI clinic or endoscopy center
* Age 18-60 years old
* Provision of written consent
* Negative upper endoscopy (oesophagogastroduodenoscopy or OGD) finding

Exclusion Criteria:

* Diabetes mellitis
* Frequent (once or more per week) acid reflux or heartburn symptoms
* Concurrent medications that affect GI motility
* Concurrent use of TCA
* History of gastric surgery
* Organic disease as cause of dyspepsia
* H. pylori infection
* Use of PPI or NSAID in the past 4 weeks
* Pregnancy
* Known hypersensitivity to PPI

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2009-12-03 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-02-19 (Actual)

PRIMARY OUTCOMES:
gastric emptying rate as measured by BreathID:Area-under-curve (AUC) values at different time points and half-emptying time (t1/2) after 8 weeks of treatment will be used as measures for gastric emptying rate | 8 weeks

SECONDARY OUTCOMES:
calorie intake in satiety test | 8 weeks
rate of adequate relief using global symptom assessment | 8 weeks
symptom scores | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Justin C.Y. Wu, MBChB(CUHK), Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong